CLINICAL TRIAL: NCT02869074
Title: Molecular and Clinical Profile of Von Willebrand Disease (VWD) in Spain (PCM-EVW-ES). Recruitment Extension, Further Data Analysis, Improvement of Registry Platform, Diagnosis and Management of VWD Application Development
Brief Title: Molecular and Clinical Profile of Von Willebrand Disease in Spain
Acronym: PCM-EVW-ES
Status: Completed | Type: Observational
Sponsor: Spanish Society of Thrombosis and Haemostasis (Other)
Collaborators: Francisco Vidal Pérez (Unknown); Maria Fernanda López Fernández (Unknown); Almudena Pérez Rodríguez (Unknown); Irene Corrales Insa (Unknown); Ana Rosa Cid Haro (Unknown)
Responsible Party: Principal Investigator, Francisco Javier Batlle Fonrodona, Senior Researcher INIBIC. A Coruña. SPAIN, Spanish Society of Thrombosis and Haemostasis
Other Study IDs: PCM-EVW-ES.SPANISH REGISTRY
Record Dates: First submitted 2016-07-29; First posted 2016-08-16 (Estimated); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Von Willebrand Disease
Keywords: von Willebrand disease (VWD); von Willebrand factor (VWF); von Willebrand factor gene; next generation sequencing; diagnosis; VWD Spanish Cohort
MeSH Terms: conditions — von Willebrand Diseases; Disease | interventions — von Willebrand Factor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Biospecimen Retention: Samples With DNA — EDTA-Blood 5 mL Citrated Blood 5 mL
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- VWD Spanish Cohort: Patients with previously diadnosis of VWD from approximately 38-40 different centers from Spain.
  Samples from these patients will be analyzed locally, and also centrally for VWF and VWFgene
  Interventions: Genetic: VWF gene analysis

INTERVENTIONS:
Genetic: VWF gene analysis — 52 exons adjacent intronic regions and promotor of VWF will be analyzed

SUMMARY:
The present Project is a third phase of the previous PCM-EVW-ES Project (Batlle et al. Thromb & Haemost 2015) with the aim of its extension, further analysis with an innovation development in the field of von Willebrand disease (VWD) based in the newer recently available methodologies. The aim of this project is to help the physician in a more uniform characterization and therapy of VWD in clinical practice, at an international level. A reduction of the expenses in the diagnosis process by using the new methodologies is pursued.

DETAILED DESCRIPTION:
The present Project is a third phase of the previous PCM-EVW-ES Project (Batlle et al. Thromb & Haemost 2015) with the aim of its extension, further analysis with an innovation development in the field of von Willebrand disease (VWD) based in the newer recently available methodologies. The aim of this project is to help the physician in a more uniform characterization and therapy of VWD in clinical practice, at an international level. A reduction of the expenses in the diagnosis process by using the new methodologies is pursued.

The specific objectives and corresponding tasks of the present project are as follows:

1. Extension of the central phenotypic and next generation sequencing (NGS) genotypic characterization of the VWD in Spain, through the prospective recruitment in the Spanish VWD cohort of approximately 500 new patients with local historical VWD diagnosis (from approximately 38 centres).

i. Improvement of the registry portal and database. ii. Recruitment criteria, phenotypic and genetic analysis of new recruited patients. In silico studies of novel von Willebrand factor gene (VWF) mutations iii. Analysis/investigation of the potential interrelationship between different clinical, phenotypic and genetic variations of the all recruited patients. iv. Validation/confirmation of the PCM-EVW-ES of the new initial diagnostic proposed algorithm including VWF NGS analysis. This project involves leading innovation and translational research with a direct impact on the quality of clinical care (applicability). To our knowledge there is no similar project in this field. Potential patents may derive from this project. It involves also development of e-learning and new information technologies (debates forum, ads, google search engine). This project may promote international collaboration.

Development of an algorithmic platform that facilitates diagnosis and therapy orientation of VWD in clinical practice using the selected data from the overwhelming amount of information that new technologies, such as NGS, are producing.

ELIGIBILITY:
Inclusion Criteria: One or more of the following:

1. VWF ≤ 30 IU/d, in 2 or more occasions.
2. Presence of multimeric abnormalities.
3. If isolated FVIII deficiency demonstration of decreased FVIII binding.
4. Presence of some VWF mutation.
5. ↑ RIPA at low concentrations of ristocetin.

Exclusion Criteria:

1. Presence of any data suggesting AVWS.
2. Absence of a signed patient informed consent

Ages: 2 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Up to 676 new patients (not previously recruited for the Spanish Registry) locally diagnosed of VWD.
Sampling Method: Non-Probability Sample
Enrollment: 790 (Actual)
Dates: Start 2017-10-03 (Actual); Primary Completion 2021-09-25 (Actual); Study Completion 2021-09-25 (Actual)

PRIMARY OUTCOMES:
Central diagnosis of 400 new VWD Spanish patients | January 2019
  Phenotype and genetic central diagnosis of 400 new VWD Spanish patients. With determinations in samples obtained after patients recruitment, VWF NGS sequencing carried out in all patients, for exons 1 to 52, adjacent intronic regions and aproximately 1300 bp of promotor region.
  A pheno-genotype will be made With a final diagnosis assignment Evaluation of pheno/genotype congruence

SECONDARY OUTCOMES:
PCM-EVW-ES project algorithm validation/confirmation | January 2019
  Evaluation of the algorithm with data from the Spanish Registry patients. Mutation results will be used in the first line of VWD diagnosis Correlation between mutations and phenotype
Potential collaboration with the International Society on Thrombosis and Haemostasis | January 2019
  Proposal for evaluation of the PCM-EVW-ES algorithm with data from other international VWD patients cohorts

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Javier BATLLE, PhD, MD, Study Chair — Complexo Hospitalario Universitario A Coruña. INIBIC. A Coruña. Spain
Locations (1):
- Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias, Spain

REFERENCES:
- [Background] Lillicrap D. von Willebrand disease: advances in pathogenetic understanding, diagnosis, and therapy. Hematology Am Soc Hematol Educ Program. 2013;2013:254-60. doi: 10.1182/asheducation-2013.1.254. PMID 24319188
- [Result] Batlle J, Perez-Rodriguez A, Corrales I, Lopez-Fernandez MF, Rodriguez-Trillo A, Loures E, Cid AR, Bonanad S, Cabrera N, Moret A, Parra R, Mingot-Castellano ME, Balda I, Altisent C, Perez-Montes R, Fisac RM, Iruin G, Herrero S, Soto I, de Rueda B, Jimenez-Yuste V, Alonso N, Vilarino D, Arija O, Campos R, Paloma MJ, Bermejo N, Toll T, Mateo J, Arribalzaga K, Marco P, Palomo A, Sarmiento L, Inigo B, Nieto Mdel M, Vidal R, Martinez MP, Aguinaco R, Cesar JM, Ferreiro M, Garcia-Frade J, Rodriguez-Huerta AM, Cuesta J, Rodriguez-Gonzalez R, Garcia-Candel F, Cornudella R, Aguilar C, Borras N, Vidal F. Molecular and clinical profile of von Willebrand disease in Spain (PCM-EVW-ES): Proposal for a new diagnostic paradigm. Thromb Haemost. 2016 Jan;115(1):40-50. doi: 10.1160/TH15-04-0282. Epub 2015 Aug 6. PMID 26245874
- [Result] Batlle J, Perez-Rodriguez A, Pinto JC, Fraga EL, Rodriguez-Trillo Tch A, Fernanda Lopez-Fernandez M. Diagnosis and management of von Willebrand disease in Spain. Semin Thromb Hemost. 2011 Jul;37(5):503-10. doi: 10.1055/s-0031-1281036. Epub 2011 Nov 18. PMID 22102193
- [Result] Goodeve A, Eikenboom J, Castaman G, Rodeghiero F, Federici AB, Batlle J, Meyer D, Mazurier C, Goudemand J, Schneppenheim R, Budde U, Ingerslev J, Habart D, Vorlova Z, Holmberg L, Lethagen S, Pasi J, Hill F, Hashemi Soteh M, Baronciani L, Hallden C, Guilliatt A, Lester W, Peake I. Phenotype and genotype of a cohort of families historically diagnosed with type 1 von Willebrand disease in the European study, Molecular and Clinical Markers for the Diagnosis and Management of Type 1 von Willebrand Disease (MCMDM-1VWD). Blood. 2007 Jan 1;109(1):112-21. doi: 10.1182/blood-2006-05-020784. Epub 2006 Sep 19. PMID 16985174
- [Result] Hashemi Soteh M, Peake IR, Marsden L, Anson J, Batlle J, Meyer D, Fressinaud E, Mazurier C, Goudemand J, Eikenboom J, Goodeve A; MCMDM-1VWD Study Group. Mutational analysis of the von Willebrand factor gene in type 1 von Willebrand disease using conformation sensitive gel electrophoresis: a comparison of fluorescent and manual techniques. Haematologica. 2007 Apr;92(4):550-3. doi: 10.3324/haematol.10606. PMID 17488667
- [Result] Budde U, Schneppenheim R, Eikenboom J, Goodeve A, Will K, Drewke E, Castaman G, Rodeghiero F, Federici AB, Batlle J, Perez A, Meyer D, Mazurier C, Goudemand J, Ingerslev J, Habart D, Vorlova Z, Holmberg L, Lethagen S, Pasi J, Hill F, Peake I. Detailed von Willebrand factor multimer analysis in patients with von Willebrand disease in the European study, molecular and clinical markers for the diagnosis and management of type 1 von Willebrand disease (MCMDM-1VWD). J Thromb Haemost. 2008 May;6(5):762-71. doi: 10.1111/j.1538-7836.2008.02945.x. Epub 2008 Mar 1. PMID 18315556
- [Result] Haberichter SL, Castaman G, Budde U, Peake I, Goodeve A, Rodeghiero F, Federici AB, Batlle J, Meyer D, Mazurier C, Goudemand J, Eikenboom J, Schneppenheim R, Ingerslev J, Vorlova Z, Habart D, Holmberg L, Lethagen S, Pasi J, Hill FG, Montgomery RR. Identification of type 1 von Willebrand disease patients with reduced von Willebrand factor survival by assay of the VWF propeptide in the European study: molecular and clinical markers for the diagnosis and management of type 1 VWD (MCMDM-1VWD). Blood. 2008 May 15;111(10):4979-85. doi: 10.1182/blood-2007-09-110940. Epub 2008 Mar 14. PMID 18344424
- [Result] Costa-Pinto J, Perez-Rodriguez A, del C Gomez-del-Castillo M, Loures E, Rodriguez-Trillo A, Batlle J, Lopez-Fernandez MF. Diagnosis of inherited von Willebrand disease: comparison of two methodologies and analysis of the discrepancies. Haemophilia. 2014 Jul;20(4):559-67. doi: 10.1111/hae.12380. PMID 25077350
- [Result] Batlle J, Lopez-Fernandez MF, Fraga EL, Trillo AR, Perez-Rodriguez MA. Von Willebrand factor/factor VIII concentrates in the treatment of von Willebrand disease. Blood Coagul Fibrinolysis. 2009 Mar;20(2):89-100. doi: 10.1097/MBC.0b013e3283254570. PMID 19786936
- [Result] Eikenboom J, Hilbert L, Ribba AS, Hommais A, Habart D, Messenger S, Al-Buhairan A, Guilliatt A, Lester W, Mazurier C, Meyer D, Fressinaud E, Budde U, Will K, Schneppenheim R, Obser T, Marggraf O, Eckert E, Castaman G, Rodeghiero F, Federici AB, Batlle J, Goudemand J, Ingerslev J, Lethagen S, Hill F, Peake I, Goodeve A. Expression of 14 von Willebrand factor mutations identified in patients with type 1 von Willebrand disease from the MCMDM-1VWD study. J Thromb Haemost. 2009 Aug;7(8):1304-12. doi: 10.1111/j.1538-7836.2009.03486.x. Epub 2009 Jun 30. PMID 19566550
- [Result] Eikenboom J, Van Marion V, Putter H, Goodeve A, Rodeghiero F, Castaman G, Federici AB, Batlle J, Meyer D, Mazurier C, Goudemand J, Schneppenheim R, Budde U, Ingerslev J, Vorlova Z, Habart D, Holmberg L, Lethagen S, Pasi J, Hill F, Peake I. Linkage analysis in families diagnosed with type 1 von Willebrand disease in the European study, molecular and clinical markers for the diagnosis and management of type 1 VWD. J Thromb Haemost. 2006 Apr;4(4):774-82. doi: 10.1111/j.1538-7836.2006.01823.x. PMID 16634746
- [Result] Tosetto A, Rodeghiero F, Castaman G, Goodeve A, Federici AB, Batlle J, Meyer D, Fressinaud E, Mazurier C, Goudemand J, Eikenboom J, Schneppenheim R, Budde U, Ingerslev J, Vorlova Z, Habart D, Holmberg L, Lethagen S, Pasi J, Hill F, Peake I. A quantitative analysis of bleeding symptoms in type 1 von Willebrand disease: results from a multicenter European study (MCMDM-1 VWD). J Thromb Haemost. 2006 Apr;4(4):766-73. doi: 10.1111/j.1538-7836.2006.01847.x. PMID 16634745
- [Result] Rodeghiero F, Castaman G, Tosetto A, Batlle J, Baudo F, Cappelletti A, Casana P, De Bosch N, Eikenboom JC, Federici AB, Lethagen S, Linari S, Srivastava A. The discriminant power of bleeding history for the diagnosis of type 1 von Willebrand disease: an international, multicenter study. J Thromb Haemost. 2005 Dec;3(12):2619-26. doi: 10.1111/j.1538-7836.2005.01663.x. PMID 16359502
- [Result] Penas N, Perez-Rodriguez A, Torea JH, Loures E, Noya MS, Lopez-Fernandez MF, Batlle J. von Willebrand disease R1374C: type 2A or 2M? A challenge to the revised classification. High frequency in the northwest of Spain (Galicia). Am J Hematol. 2005 Nov;80(3):188-96. doi: 10.1002/ajh.20470. PMID 16247740
- [Result] Corrales I, Ramirez L, Altisent C, Parra R, Vidal F. The study of the effect of splicing mutations in von Willebrand factor using RNA isolated from patients' platelets and leukocytes. J Thromb Haemost. 2011 Apr;9(4):679-88. doi: 10.1111/j.1538-7836.2011.04204.x. PMID 21251206
- [Result] Corrales I, Ramirez L, Ayats J, Altisent C, Parra R, Vidal F. Integration of molecular and clinical data of 40 unrelated von Willebrand Disease families in a Spanish locus-specific mutation database: first release including 58 mutations. Haematologica. 2010 Nov;95(11):1982-4. doi: 10.3324/haematol.2010.028977. Epub 2010 Aug 26. No abstract available. PMID 20801902
- [Result] Corrales I, Ramirez L, Altisent C, Parra R, Vidal F. Rapid molecular diagnosis of von Willebrand disease by direct sequencing. Detection of 12 novel putative mutations in VWF gene. Thromb Haemost. 2009 Mar;101(3):570-6. doi: 10.1160/th08-08-0500. PMID 19277422
- [Result] Tosetto A, Rodeghiero F, Castaman G, Goodeve A, Federici AB, Batlle J, Meyer D, Goudemand J, Eikenboom J, Schneppenheim R, Budde U, Ingerslev J, Lethagen S, Hill FG, Peake I. A comparison between two semi-quantitative bleeding scales for the diagnosis and assessment of bleeding severity in type 1 von Willebrand disease. Haemophilia. 2011 Jan;17(1):165-6. doi: 10.1111/j.1365-2516.2010.02381.x. No abstract available. PMID 21199188
- [Result] Castaman G, Goodeve A, Eikenboom J; European Group on von Willebrand Disease. Principles of care for the diagnosis and treatment of von Willebrand disease. Haematologica. 2013 May;98(5):667-74. doi: 10.3324/haematol.2012.077263. PMID 23633542
- [Result] Eikenboom J, Federici AB, Dirven RJ, Castaman G, Rodeghiero F, Budde U, Schneppenheim R, Batlle J, Canciani MT, Goudemand J, Peake I, Goodeve A; MCMDM-1VWD Study Group. VWF propeptide and ratios between VWF, VWF propeptide, and FVIII in the characterization of type 1 von Willebrand disease. Blood. 2013 Mar 21;121(12):2336-9. doi: 10.1182/blood-2012-09-455089. Epub 2013 Jan 24. PMID 23349392
- [Result] Mancuso DJ, Tuley EA, Westfield LA, Worrall NK, Shelton-Inloes BB, Sorace JM, Alevy YG, Sadler JE. Structure of the gene for human von Willebrand factor. J Biol Chem. 1989 Nov 25;264(33):19514-27. PMID 2584182
- [Result] Sadler JE, Budde U, Eikenboom JC, Favaloro EJ, Hill FG, Holmberg L, Ingerslev J, Lee CA, Lillicrap D, Mannucci PM, Mazurier C, Meyer D, Nichols WL, Nishino M, Peake IR, Rodeghiero F, Schneppenheim R, Ruggeri ZM, Srivastava A, Montgomery RR, Federici AB; Working Party on von Willebrand Disease Classification. Update on the pathophysiology and classification of von Willebrand disease: a report of the Subcommittee on von Willebrand Factor. J Thromb Haemost. 2006 Oct;4(10):2103-14. doi: 10.1111/j.1538-7836.2006.02146.x. Epub 2006 Aug 2. PMID 16889557
- [Result] Bellissimo DB, Christopherson PA, Flood VH, Gill JC, Friedman KD, Haberichter SL, Shapiro AD, Abshire TC, Leissinger C, Hoots WK, Lusher JM, Ragni MV, Montgomery RR. VWF mutations and new sequence variations identified in healthy controls are more frequent in the African-American population. Blood. 2012 Mar 1;119(9):2135-40. doi: 10.1182/blood-2011-10-384610. Epub 2011 Dec 23. PMID 22197721
- [Result] Flood VH, Gill JC, Christopherson PA, Bellissimo DB, Friedman KD, Haberichter SL, Lentz SR, Montgomery RR. Critical von Willebrand factor A1 domain residues influence type VI collagen binding. J Thromb Haemost. 2012 Jul;10(7):1417-24. doi: 10.1111/j.1538-7836.2012.04746.x. PMID 22507569
- [Result] Borras N, Batlle J, Perez-Rodriguez A, Lopez-Fernandez MF, Rodriguez-Trillo A, Loures E, Cid AR, Bonanad S, Cabrera N, Moret A, Parra R, Mingot-Castellano ME, Balda I, Altisent C, Perez-Montes R, Fisac RM, Iruin G, Herrero S, Soto I, de Rueda B, Jimenez-Yuste V, Alonso N, Vilarino D, Arija O, Campos R, Paloma MJ, Bermejo N, Berrueco R, Mateo J, Arribalzaga K, Marco P, Palomo A, Sarmiento L, Inigo B, Nieto MDM, Vidal R, Martinez MP, Aguinaco R, Cesar JM, Ferreiro M, Garcia-Frade J, Rodriguez-Huerta AM, Cuesta J, Rodriguez-Gonzalez R, Garcia-Candel F, Cornudella R, Aguilar C, Vidal F, Corrales I. Molecular and clinical profile of von Willebrand disease in Spain (PCM-EVW-ES): comprehensive genetic analysis by next-generation sequencing of 480 patients. Haematologica. 2017 Dec;102(12):2005-2014. doi: 10.3324/haematol.2017.168765. Epub 2017 Sep 29. PMID 28971901
- [Result] Perez-Rodriguez A, Batlle J, Corrales I, Borras N, Rodriguez-Trillo A, Loures E, Cid AR, Bonanad S, Cabrera N, Moret A, Parra R, Mingot-Castellano ME, Navarro N, Altisent C, Perez-Montes R, Marcellini S, Moreto A, Herrero S, Soto I, Fernandez Mosteirin N, Jimenez-Yuste V, Alonso N, de Andres Jacob A, Fontanes E, Campos R, Paloma MJ, Bermejo N, Berrueco R, Mateo J, Arribalzaga K, Marco P, Palomo A, Castro Quismondo N, Inigo B, Nieto MDM, Vidal R, Martinez MP, Aguinaco R, Tenorio M, Ferreiro M, Garcia-Frade J, Rodriguez-Huerta AM, Cuesta J, Rodriguez-Gonzalez R, Garcia-Candel F, Dobon M, Aguilar C, Batlle F, Vidal F, Lopez-Fernandez MF. Role of multimeric analysis of von Willebrand factor (VWF) in von Willebrand disease (VWD) diagnosis: Lessons from the PCM-EVW-ES Spanish project. PLoS One. 2018 Jun 20;13(6):e0197876. doi: 10.1371/journal.pone.0197876. eCollection 2018. PMID 29924855
- [Result] Borras N, Orriols G, Batlle J, Perez-Rodriguez A, Fidalgo T, Martinho P, Lopez-Fernandez MF, Rodriguez-Trillo A, Loures E, Parra R, Altisent C, Cid AR, Bonanad S, Cabrera N, Moret A, Mingot-Castellano ME, Navarro N, Perez-Montes R, Marcellin S, Moreto A, Herrero S, Soto I, Fernandez-Mosteirin N, Jimenez-Yuste V, Alonso N, de Andres-Jacob A, Fontanes E, Campos R, Paloma MJ, Bermejo N, Berrueco R, Mateo J, Arribalzaga K, Marco P, Palomo A, Quismondo NC, Inigo B, Nieto MDM, Vidal R, Martinez MP, Aguinaco R, Tenorio JM, Ferreiro M, Garcia-Frade J, Rodriguez-Huerta AM, Cuesta J, Rodriguez-Gonzalez R, Garcia-Candel F, Dobon M, Aguilar C, Vidal F, Corrales I. Unraveling the effect of silent, intronic and missense mutations on VWF splicing: contribution of next generation sequencing in the study of mRNA. Haematologica. 2019 Mar;104(3):587-598. doi: 10.3324/haematol.2018.203166. Epub 2018 Oct 25. PMID 30361419
- [Result] Batlle J, Perez-Rodriguez A, Corrales I, Borras N, Costa Pinto J, Lopez-Fernandez MF, Vidal F; PCM-EVW-ES Investigators Team. Update on Molecular Testing in von Willebrand Disease. Semin Thromb Hemost. 2019 Oct;45(7):708-719. doi: 10.1055/s-0039-1679922. Epub 2019 Apr 30. PMID 31041796
- [Result] Borras N, Garcia-Martinez I, Batlle J, Perez-Rodriguez A, Parra R, Altisent C, Lopez-Fernandez MF, Costa Pinto J, Batlle-Lopez F, Cid AR, Bonanad S, Cabrera N, Moret A, Mingot-Castellano ME, Navarro N, Perez-Montes R, Marcellini S, Moreto A, Herrero S, Soto I, Fernandez-Mosteirin N, Jimenez-Yuste V, Alonso N, de Andres-Jacob A, Fontanes E, Campos R, Paloma MJ, Bermejo N, Berrueco R, Mateo J, Arribalzaga K, Marco P, Palomo A, Castro Quismondo N, Inigo B, Del Mar Nieto M, Vidal R, Martinez MP, Aguinaco R, Tenorio M, Ferreiro M, Garcia-Frade J, Rodriguez-Huerta AM, Cuesta J, Rodriguez-Gonzalez R, Garcia-Candel F, Dobon M, Aguilar C, Corrales I, Vidal F. Unraveling the Influence of Common von Willebrand factor variants on von Willebrand Disease Phenotype: An Exploratory Study on the Molecular and Clinical Profile of von Willebrand Disease in Spain Cohort. Thromb Haemost. 2020 Mar;120(3):437-448. doi: 10.1055/s-0040-1702227. Epub 2020 Mar 5. PMID 32135566

DOCUMENTS (1):
  • Study Protocol (2016-03-31): https://cdn.clinicaltrials.gov/large-docs/74/NCT02869074/Prot_000.pdf